CLINICAL TRIAL: NCT02290639
Title: Brief Cognitive Behavioral Treatment of Deployment-Related PTSD Symptoms in Primary Care Settings: A Randomized Controlled Trial
Brief Title: Brief Cognitive Behavioral Treatment of Deployment-Related PTSD Symptoms in Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: San Antonio Military Medical Center (U.S. Federal Agency); 59th Medical Wing (U.S. Federal Agency); Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20130057H; C.2012.184d (Other: BAMC Institutional Review Board); W81XWH-08-2-0109 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Posttraumatic Stress; Posttraumatic Stress Disorder; Military; Primary Care; Cognitive Behavioral Therapy; Prolonged Exposure; Cognitive Processing Therapy; Behavioral Health Optimization Program; Behavioral Health Consultant
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Treatment (Experimental): Four 30-minute sessions of Brief Cognitive Behavioral treatment starting immediately upon randomization.
  Interventions: Behavioral: Brief Cognitive Behavioral Treatment
- Minimal Contact followed by treatment (Active Comparator): 6-week Minimal Contact period consisting of weekly phone calls starting immediately upon randomization. Experimental treatment will be provided to all subjects upon completion of Minimal Contact period.
  Interventions: Behavioral: Brief Cognitive Behavioral Treatment; Behavioral: Minimal Contact

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Treatment — Cognitive-behavioral therapy (CBT) protocol designed specifically for use by behavioral health consultants (BHC) working in an integrated primary care setting. The treatment will be provided by a BHC in four 30-minute appointments scheduled approximately once a week in primary care over a one month period. Treatment content was largely drawn from a Prolonged Exposure model, but also includes elements of Cognitive Processing Therapy.
Behavioral: Minimal Contact — Participants assigned to minimal contact (MC) will be asked to not work with another therapist or seek additional treatment for trauma-related difficulties during the 6-week MC period. They will be called once per week by the Behavioral Health Consultant (BHC) in order to monitor their status and to provide support as needed. The calls will be limited to 5-10 minutes.
  Arms: Minimal Contact followed by treatment

SUMMARY:
A significant number of veterans of the wars in Iraq and Afghanistan are affected by posttraumatic stress disorder (PTSD). The limited reach of effective treatments for PTSD into the veteran population is at least partially due to the perceived stigma by service members for seeking help in traditional specialty mental health clinics. A comprehensive approach to PTSD treatment in a veteran population should provide alternative sources for accessing effective psychotherapy treatments. The purpose of study is to conduct a randomized clinical trial comparing a brief (four 30-minute sessions delivered over 6 weeks) cognitive-behavioral therapy (CBT) protocol designed specifically for use by behavioral health consultants working in an integrated primary care setting to a minimal contact 6-week control. The primary outcome measure is PTSD symptom relief.

DETAILED DESCRIPTION:
A significant number of veterans of the wars in Iraq and Afghanistan are affected by posttraumatic stress disorder (PTSD) yet relatively few are receiving evidence-based treatments (Tanielian, Jaycox, Schell, Marshall, Burnham, Eibner, et al. 2008). The limited reach of effective treatments for PTSD into the veteran population is at least partially due to the perceived stigma by service members for seeking help in traditional specialty mental health clinics (Hoge, Castro, Messer, McGurk, Cotting, & Koffman, 2004). A comprehensive approach to PTSD treatment in a veteran population should provide alternative sources for accessing effective psychotherapy treatments. This study builds upon a pilot study conducted at Brooke Army Medical Center and the Wilford Hall Medical Center (now the Wilford Hall Ambulatory Surgical Center) (C.2009.022, IRBNet 363516). Using the treatment protocol developed and found to be effective as part of this pilot, the purpose of study is to conduct a randomized clinical trial comparing a brief (four 30-minute sessions delivered over 6 weeks) cognitive-behavioral therapy (CBT) protocol designed specifically for use by behavioral health consultants working in an integrated primary care setting to a minimal contact 6-week control. Up to 75 Service Members with deployment-related PTSD symptoms will be consented, enrolled, and treated until treatment has been completed for 60. The primary outcome measure is PTSD symptom relief.

OBJECTIVES/SPECIFIC AIMS/RESEARCH QUESTIONS:

1. Will Operation Iraqi Freedom/Operation Enduring Freedom/Operation New Dawn (OIF/OEF/OND) veterans with PTSD symptoms accept an offer of cognitive behavioral therapy (CBT) treatment in the primary care setting versus a referral to specialty care?
2. Will a brief (four 30-minute appointments) CBT protocol designed for use by behavioral health consultants working in primary care significantly reduce PTSD symptom severity in OIF/OEF/OND veterans in comparison to a minimal contact condition?
3. Are there characteristics of patients at pre-treatment, e.g., demographic variables, level of co-morbid depression, that predict a relatively better or worse response to PTSD treatment in primary care?

ELIGIBILITY:
Inclusion Criteria:

1. active duty, reserve, guard, separated, or retired OIF/OEF/OND veterans seeking care in primary care for deployment-related PTSD symptoms
2. Symptomatic for PTSD will be defined as a minimum score of 32 on the PTSD CheckList -Stressor-specific (PCL-S)
3. English speaking
4. If individuals are taking psychotropic medication, a 4-week stabilization period may be required prior to enrollment, depending upon the medication, half-life, and anticipated interaction with the ability to engage in behavioral therapy

Exclusion Criteria:

1. moderate to severe suicide risk
2. current alcohol dependence, psychotic disorder, significant dissociative disorder
3. severe brain injury
4. Patients who are currently receiving talk therapy for trauma-related symptoms will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-12; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
PTSD Symptom Scale, Interview Version (PSS-I); to assess change in PTSD symptomatology and/or diagnosis from baseline to multiple follow up time points | Baseline, 2 weeks post-tx, 8 weeks post-tx, 6 months post-tx
  The PSS-I is a 20-minute, 17-item clinical interview that evaluates each of the DSM-IV PTSD symptoms during the past 2 weeks on a frequency/severity scale (Foa, Riggs, Dancu, & Rothbaum, 1993). The PSS-I is comparable to the gold standard employed in studies of veterans (the Clinician Administered PTSD Scale; CAPS) yet takes considerably less time to administer (Foa & Tolin, 2000). Each symptom is rated on a 4-point scale ranging from 0 (not at all) to 3 (very much). Subscale scores are calculated by summing items in each of the PTSD symptom clusters: re-experiencing, avoidance, and arousal. The scale has excellent internal consistency (α = .85), test-retest reliability (.80), and inter-rater reliability (kappa = .97; Foa et al, 1993). This measure will be administered by a blinded Independent Evaluator at each study site.
PTSD Checklist - Stressor-Specific Version (PCL-S); to assess change in PTSD symptomatology from baseline throughout treatment and at multiple follow up time points | Baseline, Weekly during treatment (4 time points), 2 weeks post-tx, 8 weeks post-tx, 6 months post-tx
  The PCL-S is a 17 item self-report measure based upon the PTSD Checklist - Military (PCL-M; Weathers, Litz, Herman, Huska, & Keane, 1993) that evaluates how much participants have been bothered by PTSD symptoms in the past month as a result of the stressful life events identified by either the participant, or by the Independent Evaluator following administration of the PSS-I. Each item of the PCL-S is scored on a five-point scale ranging from 1 (-not at all‖) to 5 (-extremely‖). The measure is divided into 3 subscales: Re-experiencing symptoms (items 1- 5); Avoidance/ Emotional Numbing symptoms (items 6- 12); and Hyper-arousal symptoms (items 12-17).

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Peterson, PhD, ABPP, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Wilford Hall Ambulatory Surgical Center Family Medicine Clinic, Lackland Air Force Base, Texas
  - Joint Base San Antonio, Randolph Air Force Base, Texas

REFERENCES:
- [Derived] Cigrang JA, Rauch SA, Mintz J, Brundige AR, Mitchell JA, Najera E, Litz BT, Young-McCaughan S, Roache JD, Hembree EA, Goodie JL, Sonnek SM, Peterson AL; STRONG STAR Consortium. Moving effective treatment for posttraumatic stress disorder to primary care: A randomized controlled trial with active duty military. Fam Syst Health. 2017 Dec;35(4):450-462. doi: 10.1037/fsh0000315. PMID 29283612